CLINICAL TRIAL: NCT02508805
Title: Open Randomised Comparative Study of the Efficacy and Safety of Neuromultivit (Solution for Injections, 2 ml) in Patients With Vertebrogenic Radiculopathy
Brief Title: Safety and Efficacy of Neuromultivit in Treatment of Vertebrogenic Radiculopathy
Acronym: NMRUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Valeant Russia, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NM-01RUS; 224 (Registry Identifier: registration study)
Record Dates: First submitted 2015-07-17; First posted 2015-07-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Vertebrogenic Radiculopathy L5, S1
MeSH Terms: interventions — Diclofenac; tizanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromultivit +Voltaren+Sirdalud (Experimental): Neuromultivit 2ml i.m. once a day for 7 days, then 2 ml i.m. one time every other day for 10 days.
  Voltaren 100mg per os once a day for 20 days. Sirdalud 2 mg per os three times a day for 20 days.
  Interventions: Drug: Neuromultivit; Drug: Voltaren; Drug: Sirdalud
- Voltaren+Sirdalud alone (Active Comparator): Voltaren 100mg per os once a day for 20 days Sirdalud 2 mg per os three times a day for 20 days
  Interventions: Drug: Voltaren; Drug: Sirdalud

INTERVENTIONS:
Drug: Neuromultivit
  Arms: Neuromultivit +Voltaren+Sirdalud
Drug: Voltaren
Drug: Sirdalud

SUMMARY:
The purpose of the study is to assess the efficacy and safety of Neuromultivit (solution for injections) in treatment of vertebrogenic radiculopathy L5, S1 in comparison with standard therapy. The patients are randomised into two groups: standard therapy group and standard therapy plus Neuromultivit group.

DETAILED DESCRIPTION:
Group 1 (50 patients) receive Neuromultivit (2 ml per day, i.m.) for 7 days, then -Neuromultivit (2 ml per day, i.m.) every other day for 10 days and standard therapy for 20 days.

Group 2 (50 patients) receive only standard therapy for 20 days.

Standard therapy involves:

* Voltaren (100 mg prolonged-released film-coated tablets once daily) for 20 days
* Sirdalud (2 mg tablets three times a day) for 20 days

ELIGIBILITY:
Inclusion Criteria:

* diagnosed vertebrogenic radiculopathy L5, S1
* radicular pain syndrome
* changes in the low back CT and MRI scans
* minimum 40 mm intensity of spontaneous back pain, rated on the VA scale
* 1 month exacerbation phase; nonuse of any B-group vitamins before the trial
* negative urine pregnancy test; Patient Informed Consent

Exclusion Criteria:

* tumors, inflammatory infections, any neurological diseases, imitating the symptoms of radiculopathy
* concomitant life-threatening medical conditions
* simultaneous administration of acetylsalicylic acid, levodopa, prednisolone; any psychiatric diseases
* epilepsy, alcohol and drug addiction
* pregnancy and breast-feeding
* any condition preventing CT and MRI tests, including obesity and special devices
* participation in any other clinical study 1 month before enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain Intensity at Rest and with Activity in Visual Analoguе Scale | baseline and 3 weeks
  Self reported pain intensity over the last 24 hours. The amount of pain is marked on a horizontal line at a certain point which reflects pain perception best: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

SECONDARY OUTCOMES:
Change from Baseline in Pain Quality and Intensity in McGill Pain Questionnaire | baseline and 3 weeks
  Self reported quality and intensity of pain, described by selecting 7 words, which reflect pain perception best, from 20 groups: three words from groups 1-10, two words from groups 11-15, a single word from group 16, one word from groups 17-20.
Change from Baseline in Low Back Pain Intensity in Aberdeen Back Pain Scale | baseline and 3 weeks
  Self reported effect of pain on body functions and daily activities. The scores of responses to 19 questions (6 multiple choice questions and 13 single choice questions) are summed, yielding a total between 0 and 100 with higher values representing greater disability.
Change from Baseline in Low Back Pain Intensity in Quebec Back Pain Disability Scale | baseline and 3 weeks
  Self reported pain related functional limitations to 20 activities. The degree of difficulty in performing these daily activities is scored from 0-5 (0 = no effort, 5 = not able to), yielding a total between 0 and 100 with higher values representing greater disability.

OTHER OUTCOMES:
Change from Baseline in Systolic Blood Pressure at 10 Days | baseline and 10 days
Change from Baseline in Systolic Blood Pressure at 3 weeks | baseline and 3 weeks
Change from Baseline in Heart Rate and Rhythm (Electrocardiogram) at 3 weeks | baseline and 3 weeks
Change from Baseline in Full Blood Count at 3 weeks | baseline and 3 weeks
Change from Baseline in Urine Test at 3 weeks | baseline and 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Farit Khabirov, MD, DSc, Prof, Principal Investigator — State Autonomous Institution Republican Clinical Centre of Neurology
Locations (1):
- State Autonomous Institution Republican Clinical Centre of Neurology, Kazan', Tatarstan Republic, Russia